CLINICAL TRIAL: NCT03343704
Title: A Phase III, Case Series Clinical Study of the Reversal of the Anticoagulant Effects of Dabigatran by Intravenous Administration of Idarucizumab (BI 655075) in Patients Treated With Dabigatran Etexilate Who Have Uncontrolled Bleeding or Require Emergency Surgery or Procedures.
Brief Title: This Study Looks at the Effects of Idarucizumab in Patients Who Take Dabigatran and Need Emergency Surgery or Are Bleeding
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1321-0019
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Results first posted 2021-08-20 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — idarucizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - patients with uncontrolled or life-threatening bleeding (Experimental)
  Interventions: Drug: Idarucizumab
- Group B - patients not bleeding but requiring emergency surgery or invasive procedure (Experimental)
  Interventions: Drug: Idarucizumab

INTERVENTIONS:
Drug: Idarucizumab — Intravenous
  Other Names: PRAXBIND, Praxbind, Prizbind

SUMMARY:
The primary objective is to demonstrate reversal of the anticoagulant effect of dabigatran in patients treated with dabigatran etexilate who have uncontrolled or life-threatening bleeding requiring urgent intervention, and in patients treated with dabigatran etexilate who require emergency surgery or other invasive procedure.

The secondary objectives are to assess the reduction or cessation of bleeding, evaluate the clinical outcomes, safety and the pharmacokinetics of dabigatran in the presence of idarucizumab.

ELIGIBILITY:
Inclusion criteria:

* ≥ 18 years at screening.
* Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Currently taking dabigatran etexilate
* They meet the following criteria:

  * Group A: Overt bleeding judged by the physician to require a reversal agent. OR
  * Group B: A condition requiring emergency surgery or invasive procedure where adequate hemostasis is required. Emergency is defined as within the following 8 hours.

Exclusion criteria:

Group A:

* Patients with minor bleeding (e.g. epistaxis, hematuria) who can be managed with standard supportive care.
* Patients with no clinical signs of bleeding.
* Contraindications to study medication including known hypersensitivity to the drug or its excipients (subjects with hereditary fructose intolerance may react to sorbitol).

Group B:

* A surgery or procedure which is elective or where the risk of uncontrolled or unmanageable bleeding is low.
* Contraindications to study medication including known hypersensitivity to the drug or its excipients (subjects with hereditary fructose intolerance may react to sorbitol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - Beijing AnZhen Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Cardiovascular Institute and Fu Wai Hospital, Beijing
  - First Affiliated Hospital of Dalian Medical University, Dalian
  - Guangdong Provincial People's Hospital, Guangzhou
  - Sun yet-sen Memorial Hospital, Sun yet-sen Univesity, Guangzhou
  - 2nd Affiliated Hosp Zhejiang University College of Medical, Hangzhou
  - Zhejiang Province People's Hospital, Hangzhou
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing, Jiangsu Province
  - Shanghai First People's Hospital, Shanghai
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi
  - The First Affiliated Hospital of Wenzhou Med College, Wenzhou

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was to demonstrate the reversal of the anticoagulant effects of dabigatran by intravenous administration of idarucizumab in patients treated with dabigatran etexilate who had uncontrolled bleeding or required emergency surgery or procedures over treatment period of 1 day following by 30 days follow-up.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Group A - Patients With Uncontrolled or Life-threatening Bleeding: Two vials of 2.5 grams (g) of idarucizumab (BI 655075) (Total: 5g) were administered via intravenous infusions once over a 1-day treatment period. Two vials of idarucizumab were administered no more than 15 minutes apart.
  Patients who were taking dabigatran etexilate and had uncontrolled or life-threatening bleeding requiring urgent medical or surgical intervention were included in this group.
- Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure: Two vials of 2.5 grams (g) of idarucizumab (BI 655075) (Total: 5g) were administered via intravenous infusions once over a 1-day treatment period. Two vials of idarucizumab were administered no more than 15 minutes apart.
  Patients included in this group were those who were taking dabigatran etexilate and may not be bleeding, but do require an emergency surgery or other invasive procedure for a condition other than bleeding, where therapeutic anticoagulation with dabigatran etexilate was undesirable.
Period: Overall Study
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Started | 13 | 6
Completed | 12 | 4
Not Completed | 1 | 2
Not completed — Refused to complete follow up | 0 | 1
Not completed — Death | 0 | 1
Not completed — Reluctant to collect blood and received telephone follow up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): include all patients who are administered with idarucizumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure | Total
Number analyzed (Participants) | 13 | 6 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.4 (12.3) | 62.8 (10.6) | 71.4 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 8 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 6 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Reversal of Anticoagulant Effect of Dabigatran Based on Central Laboratory Determination of Ecarin Clotting Time
Description: Maximum reversal of anticoagulant effect of dabigatran based on central laboratory determination of ecarin clotting time is reported.
  The maximum reversal of anticoagulant effect of dabigatran is defined for patients with at least one post-dose coagulation test results and pre-dose result higher than 100% Upper limit of normal (ULN). Maximum reversal is calculated as 100% x (pre-dose value - post-dose value)/(pre-dose value - 100% ULN). If the calculated reversal is > 100, it was set to 100. 100% ULN is 41.26 seconds.
Time Frame: From the end of first infusion up to 4 hours after the completion of the second infusion on Day 1 of the treatment period.
Population: Pharmacodynamic (PD) set (PDS): comprise all patients in the treated set who provided at least one evaluable pre-dose and at least one post-dose observation for PD endpoints or biomarker measures. Only participants with non-missing outcomes are included in the analysis.
Measure: Median (95% Confidence Interval); unit: Percentage
Groups:
- Total: All participants in Group A or B were included in this group.
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure | Total
Number analyzed (Participants) | 6 | 4 | 10
Percentage | 100.0 [100.0 to 100.0] | 100.0 [96.8 to 100.0] | 100.0 [100.0 to 100.0]

2. Primary Outcome: Maximum Reversal of Anticoagulant Effect of Dabigatran Based on Central Laboratory Determination of Diluted Thrombin Time
Description: Maximum reversal of anticoagulant effect of dabigatran based on central laboratory determination of diluted thrombin time is reported.
  The maximum reversal of anticoagulant effect of dabigatran is defined for patients with at least one post-dose coagulation test results and pre-dose result higher than 100% Upper limit of normal (ULN). Maximum reversal is calculated as 100% x (pre-dose value - post-dose value)/(pre-dose value - 100% ULN). If the calculated reversal is > 100, it was set to 100. 100% ULN is 35.54 seconds.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percentage
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure | Total
Number analyzed (Participants) | 5 | 4 | 9
Percentage | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0]

3. Secondary Outcome: Percentage of Participants Achieving Cessation of Bleeding Within 24 Hours After Completion of Second Infusion (for Group A Only)
Description: Percentage of participants achieving cessation of bleeding within 24 hours after completion of second infusion for Group A is reported.
Time Frame: Up to 24 hours after the completion of the second infusion on Day 1 of the treatment period.
Population: Treated set (TS): include all patients who are administered with idarucizumab. Patients with no evaluable post-baseline bleeding assessment are excluded. This analysis only included patients with uncontrolled or life-threatening bleeding, and non-Intracranial Hemorrhage (non-ICH) in Group A.
Measure: Number; unit: Percentage of participants
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding
Number analyzed (Participants) | 9
Percentage of participants | 55.6

4. Secondary Outcome: Number of Participants With Major Bleeding (for Group B Only) Intra-operatively and up to 24 Hours Post-surgery
Description: Number of participants with major bleeding (for Group B only) intra-operatively and up to 24 hours post-surgery per International Society for Thrombosis and Hemostasis (ISTH) classification is reported.
Time Frame: Up to 24 hours post-surgery.
Population: Treated set (TS): include all patients who are administered with idarucizumab. This analysis only included patients not bleeding but requiring emergency surgery or invasive procedure (Group B).
Measure: Count of Participants; unit: Participants
Arm/Group | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Number analyzed (Participants) | 6
Participants
  Minor | 0
  Major | 1
  Major, Life -Threatening or Fatal | 0
  Not assessable | 0

5. Secondary Outcome: Minimum Unbound Sum Dabigatran Concentrations Since the End of First Infusion up to 4 Hours After the Completion of the Last Infusion (Cmin,1)
Description: Minimum unbound sum dabigatran concentrations since the end of first infusion up to 4 hours after the completion of the last infusion (Cmin,1) is reported.
Time Frame: Just prior to the second infusion (last infusion) and 10 minutes (min), 30 min, 1 hour (h), 2 h, and 4 h after the end of the second infusion.
Population: Pharmacokinetic (PK) set (PKS): comprise all patients in the TS who provided at least one PK endpoint. The PKS will be used for all PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Number analyzed (Participants) | 6 | 4
nanogram per milliliter | 1 (0) | 1 (0)

6. Secondary Outcome: Maximum Reversal of Anticoagulation as Measured by Activated Partial Thromboplastin Time (aPTT)
Description: Maximum reversal of anticoagulation as measured by activated partial thromboplastin time (aPTT) is reported.
  The reversal of anticoagulant effect of dabigatran is defined for patients with at least one post-dose coagulation test results and pre-dose result higher than 100% Upper limit of normal (ULN). Maximum reversal is calculated as 100% x (pre-dose value - post-dose value)/(pre-dose value - 100% ULN). If the calculated reversal is > 100, it was set to 100. 100% ULN is 39.80 seconds.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percentage
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure | Total
Number analyzed (Participants) | 5 | 4 | 9
Percentage | 100 [67.9 to 100.0] | 100 [98.3 to 100.0] | 100 [98.3 to 100.0]

7. Secondary Outcome: Maximum Reversal of Anticoagulation as Measured by Thrombin Time (TT)
Description: Maximum reversal of anticoagulation as measured by thrombin time (TT) is reported.
  The reversal of anticoagulant effect of dabigatran is defined for patients with at least one post-dose coagulation test results and pre-dose result higher than 100% Upper limit of normal (ULN). Maximum reversal is calculated as 100% x (pre-dose value - post-dose value)/(pre-dose value - 100% ULN). If calculated reversal is > 100, it was set to 100. 100% ULN is 14.22 seconds.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percentage
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure | Total
Number analyzed (Participants) | 6 | 4 | 10
Percentage | 100 [100.0 to 100.0] | 100 [100.0 to 100.0] | 100 [100.0 to 100.0]

8. Secondary Outcome: Numbers of Participants With Any Adverse Events - on Treatment
Description: Numbers of participants with any adverse events during on treatment period is reported.
Time Frame: Since the first infusion up until 5 days after the completion of the second infusion.
Population: Treated set (TS): include all patients who are administered with idarucizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Number analyzed (Participants) | 13 | 6
Participants | 11 | 6

9. Secondary Outcome: Numbers of Participants With Any Adverse Events - Including Post Treatment Period
Description: Numbers of participants with any adverse events until end of study is reported.
Time Frame: Since informed consent up to 30 days (± 7 days) after the completion of the second infusion, up to 37 days.
Population: Treated set (TS): include all patients who are administered with idarucizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Number analyzed (Participants) | 13 | 6
Participants | 13 | 6

10. Secondary Outcome: Number of Participants With Serious Adverse Events - on Treatment
Description: Number of participants with Serious adverse events during on treatment period is reported.
Time Frame: Since the first infusion up until 5 days after the completion of the second infusion.
Population: Treated set (TS): include all patients who are administered with idarucizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Number analyzed (Participants) | 13 | 6
Participants | 3 | 1

11. Secondary Outcome: Number of Participants With Serious Adverse Events - Including Post Treatment Period
Description: Number of participants with Serious adverse events until the end of study is reported.
Time Frame: Since informed consent up to 30 days (± 7 days) after the completion of the second infusion, up to 37 days.
Population: Treated set (TS): include all patients who are administered with idarucizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Number analyzed (Participants) | 13 | 6
Participants | 7 | 3

12. Secondary Outcome: Number of Participants With Drug-related Adverse Events - on Treatment
Description: Numbers of patients with drug-related adverse events during on treatment period is reported.
Time Frame: Since the first infusion up until 5 days after the completion of the second infusion.
Population: Treated set (TS): include all patients who are administered with idarucizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Number analyzed (Participants) | 13 | 6
Participants | 2 | 1

13. Secondary Outcome: Number of Participants With Drug-related Adverse Events - Including Post Treatment Period
Description: Numbers of patients with drug-related adverse events until end of study is reported.
Time Frame: Since informed consent up to 30 days (± 7 days) after the completion of the second infusion, up to 37 days.
Population: Treated set (TS): include all patients who are administered with idarucizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Number analyzed (Participants) | 13 | 6
Participants | 2 | 1

14. Secondary Outcome: Number of Participants With Immune Reaction Adverse Event - on Treatment
Description: Number of participants with immune reaction adverse event during on treatment period is reported.
Time Frame: Since the first infusion up until 5 days after the completion of the second infusion.
Population: Treated set (TS): include all patients who are administered with idarucizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Number analyzed (Participants) | 13 | 6
Participants | 3 | 0

15. Secondary Outcome: Number of Participants With Immune Reaction Adverse Event - Including Post Treatment Period
Description: Number of participants with immune reaction adverse event until end of study is reported.
Time Frame: Since informed consent up to 30 days (± 7 days) after the completion of the second infusion, up to 37 days.
Population: Treated set (TS): include all patients who are administered with idarucizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Number analyzed (Participants) | 13 | 6
Participants | 3 | 0

16. Secondary Outcome: Number of Participants With Thrombotic Events - on Treatment
Description: Number of participants with thrombotic events (ischemic stroke, myocardial infarction, pulmonary embolism, deep vein thrombosis, systemic embolism) during on treatment period is reported.
Time Frame: Since the first infusion up until 5 days after the completion of the second infusion.
Population: Treated set (TS): include all patients who are administered with idarucizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Number analyzed (Participants) | 13 | 6
Participants | 1 | 1

17. Secondary Outcome: Number of Participants With Thrombotic Events - Including Post Treatment Period
Description: Number of participants with thrombotic events (ischemic stroke, myocardial infarction, pulmonary embolism, deep vein thrombosis, systemic embolism) until end of study is reported.
Time Frame: Since informed consent up to 30 days (± 7 days) after the completion of the second infusion, up to 37 days.
Population: Treated set (TS): include all patients who are administered with idarucizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
Number analyzed (Participants) | 13 | 6
Participants | 2 | 3

ADVERSE EVENTS:
Time Frame: Since informed consent up to 30 days (± 7 days) after the completion of the second infusion, up to 37 days.
Description: Treated set (TS): include all patients who are administered with idarucizumab.
Arm/Group | Group A - Patients With Uncontrolled or Life-threatening Bleeding | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure
All-Cause Mortality (participants affected / at risk) | 0/13 | 1/6
Serious Adverse Events (participants affected / at risk) | 7/13 | 3/6
Other Adverse Events (participants affected / at risk) | 13/13 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - Patients With Uncontrolled or Life-threatening Bleeding (N=13) | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Seizure (Nervous system disorders) | 0 | 1
Thalamic infarction (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 2 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertensive urgency (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A - Patients With Uncontrolled or Life-threatening Bleeding (N=13) | Group B - Patients Not Bleeding But Requiring Emergency Surgery or Invasive Procedure (N=6)
Anaemia (Blood and lymphatic system disorders) | 3 | 3
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1
Hyperfibrinolysis (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dysbiosis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 0
Chest discomfort (General disorders) | 2 | 1
Chest pain (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 1
Anal infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 2
Pneumonia (Infections and infestations) | 2 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Anal injury (Injury, poisoning and procedural complications) | 1 | 0
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Urethral injury (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Antithrombin III decreased (Investigations) | 1 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 1
Blood cholinesterase decreased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine decreased (Investigations) | 0 | 1
Blood fibrinogen decreased (Investigations) | 0 | 1
Blood fibrinogen increased (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Blood uric acid decreased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Fibrin D dimer increased (Investigations) | 2 | 1
Fibrin degradation products increased (Investigations) | 1 | 1
Gamma-glutamyltransferase decreased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
High density lipoprotein decreased (Investigations) | 0 | 1
Lymphocyte percentage decreased (Investigations) | 0 | 1
Monocyte percentage decreased (Investigations) | 0 | 1
Myoglobin blood increased (Investigations) | 0 | 1
Neutrophil percentage increased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 1 | 0
Pulmonary arterial pressure increased (Investigations) | 1 | 0
Thrombin time prolonged (Investigations) | 1 | 1
Troponin I increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 2 | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT03343704/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT03343704/SAP_001.pdf